CLINICAL TRIAL: NCT06644937
Title: Single-arm Clinical Trial of TACE in Combination With Icaritin as Adjuvant Therapy After Surgery in Patients With Hepatocellular Carcinoma at High Risk of Recurrence
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-281-01
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: hepatocellular carcinoma; RFS; adjuvant therapy after surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE combination with icaritin (Experimental)
  Interventions: Drug: TACE combined with Acoradine

INTERVENTIONS:
Drug: TACE combined with Acoradine — Transcatheter hepatic arterial chemoembolization (TACE) : the treatment interval was 28 days, the window period was ± 7 days. Subjects received a maximum of 4 TACE treatments; reduced and delayed treatment: laboratory tests were performed before the start of each cycle of TACE, with investigator criteria confirming whether TACE treatment was feasible.
  Acoradine: 6 tablets bid, taken after meals for 6 months or until intolerable or progressive disease (starting one month after surgery) .

SUMMARY:
To assess 1-year recurrence-free survival (RFS) in patients with hepatocellular carcinoma (HCC) who are at high risk of Inguinal orchiectomy recurrence usingTACE combined with icaritin

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily cooperated with the study and signed the informed consent,
2. Male or female, 18 years old ≤ age ≤75 years old,
3. The histopathologic diagnosis was hepatocellular carcinoma
4. R0 resection was performed within 4 to 8 weeks before recruitment (patients who were confirmed to have R0 resection by imaging and pathological examination were excluded from the study group if the residual R1, residual R2 or the margin of resection were not clear)
5. To satisfy any of the following high risk factors for postoperative recurrence of hepatocellular carcinoma:

   I) BCLC stage B (> 3 tumors, regardless of size or number, at least one of which is > 3 cm in diameter) ; ii) single tumor ≥5 cm in diameter; III) intraoperative or postoperative pathological findings of vascular invasion (including microvascular invasion and VP1/VP2 portal vein invasion) ; IV) histopathologic grade of low differentiation; v) capsular invasion or loss with unclear border; VI) direct invasion of adjacent organs
6. ECOG performance status score of 0-1 and Child-Pugh score of 5-6
7. None of the patients had received anti-tumor therapy for hepatocellular carcinoma, including systemic therapy and local therapy (except for 1-2 prophylactic TACE or HAIC 4-8 weeks after radical therapy) .
8. Subjects who received radical therapy, if required, were allowed to receive 1-2 prophylactic TACE/Haic treatments 4-8 weeks after surgery (on demand and not necessarily)

Exclusion Criteria:

1. Known sarcomatoid hepatocellular carcinoma/mixed hepatocellular carcinoma-cholangiocarcinoma/fibrolamellar hepatocellular carcinoma;
2. A history of other malignancies in the past 5 years or at the same time;
3. Severe functional impairment of other important organs such as heart, brain, lung and kidney;
4. Patients with a history of immunodeficiency or autoimmune disease;
5. Evidence of tumor recurrence or metastasis before enrollment;
6. Known hypersensitivity to active ingredients, excipients, or history of severe allergy to any other monoclonal antibody, anti-angiogenic drugs;
7. Patients with a history of hepatic encephalopathy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
1 year recurrence-free survival rate ,1-year RFSR. | 1 year
  1 year recurrence-free survival rate ,1-year RFSR.

SECONDARY OUTCOMES:
TTR( time to recurrence) | 1year
  TTR( time to recurrence)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China